CLINICAL TRIAL: NCT03867279
Title: Flossing Technique Together With a Protocol of Neuromuscular Reeducation Exercises in the Improvement of Dorsiflexion of the Ankle and the Perception of Effort When Performing a Squat in Trained Subjects. A Randomized Clinical Trial.
Brief Title: Flossing Technique With Neuromuscular Reeducation Exercises in Trained Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLOSSING
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Weight, Body
Keywords: Weightlifters; Flossbands; Clinical Trial; Physical Therapy; Squat
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flossing (Experimental): The subjects included in this group will perform a protocol of reeducation exercises plus the application of the Flossing technique. The intervention will last 4 weeks, with two weekly sessions of 15 minutes each
  Interventions: Other: Flossing
- Reeducation exercises (Active Comparator): The subjects included in this group will carry out a protocol of reeducation exercises. The intervention will last 4 weeks, with two weekly sessions of 15 minutes each
  Interventions: Other: Reeducation exercises

INTERVENTIONS:
Other: Flossing — The reeducation exercises are: lunge and hold (the subject performs a lunge increasing the dorsiflexion of the ankle, advancing the tibia as much as possible without taking off the heel of the floor and without valgus of the knee, 15 repetition of 10 seconds of duration each); back squat (squat with a pike supported on scapulae); and chaturanga (from the prone position with extension of elbows and spine, the subject raises upper antero iliac spines performing a shoulder flexion and raising the pelvis to the ceiling maintaining the hip flexion and knees extended and keeping the heels touching the ground. The subjects included in this group will perform the exercises while a compression band is applied to the ankle.
  Arms: Flossing
Other: Reeducation exercises — The reeducation exercises are: lunge and hold (the subject performs a lunge increasing the dorsiflexion of the ankle, advancing the tibia as much as possible without taking off the heel of the floor and without valgus of the knee, 15 repetition of 10 seconds of duration each); back squat (squat with a pike supported on scapulae); and chaturanga (from the prone position with extension of elbows and spine, the subject raises upper antero iliac spines performing a shoulder flexion and raising the pelvis to the ceiling maintaining the hip flexion and knees extended and keeping the heels touching the ground.
  Arms: Reeducation exercises

SUMMARY:
Introduction. A deficit of dorsiflexion and motor control can limit the performance of a squat. Neuromuscular reeducation exercises, mobility and elasticity are used in the neuromuscular control and mobility of the kinetic chain. The Flossing technique is applied to improve ankle mobility and the perception of effort.

Objective. To compare the efficacy of a protocol for neuromuscular reeducation exercises, mobility and elasticity, and the Flossing technique in ankle mobility and perception of effort when performing squats.

Study design. Randomized, multicenter, single-blind clinical study with a follow-up period.

Methodology. 40 weightlifters included in the study will be assigned randomly to the study groups: experimental (protocol of reeducation exercises plus the application of the Flossing technique) and control (protocol of reeducation exercises). The intervention will last 4 weeks, with two weekly sessions of 15 minutes each. The variables of the study will be the range of movement of ankle dorsiflexion (Weight Bearing Lunge Test) and the perception of the effort during the squat (Borg scale). A descriptive statistical analysis will be carried out calculating the main statistical characteristics. The distribution of the sample will be analyzed using the Kolmogorov-Smirnof test. In case of homogeneity, parametric tests will be used to calculate changes after each evaluation (t-student) and the intra- and intersubject effect (repeated measures ANOVA).

Expected results. Improvement in dorsiflexion of the ankle and decrease in the perception of effort during the squat.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 24 years old
* Male
* That they be weight lifters with at least one year of experience
* That they do not present musculoskeletal injury or pathology in the three months prior to the beginning of the study

Exclusion Criteria:

* Can not be present during the 6 weeks of the intervention and the evaluations will be excluded
* Under pharmacological treatment
* Who are performing another physiotherapy study
* Not sign the informed consent document.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline dorsal ankle flexion after treatment and at a month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The dorsal ankle flexion will be measured with the Weight-bearing lunge test. The subject will stand in front of a wall, using a tape measure that goes from the wall to the first toe. The subject will perform the greatest dorsiflexion of the ankle that allows him to touch the wall without lifting the ankle. The greater distance that this objective achieves will be the reference value. The unit of measurement of this test is the centimeter, indicating a higher score a greater range of ankle movement in dorsiflexion.

SECONDARY OUTCOMES:
Change from baseline level of effort perceived after treatment and at a month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The level of effort will be measured with the modified Borg scale. With this test, the level of effort perceived by the athlete when performing the gesture of the squat will be measured. With the subject standing you will be asked to perform a squat, asking him to indicate on the scale what his level of effort has been. This scale has a range of 0 to 10 points (where 0 indicates the minimum degree of effort, and 10 the maximum effort referred by the subject).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain